CLINICAL TRIAL: NCT02437513
Title: NewBreez for Airway Protection in Head and Neck Cancer Patients With Chronic Aspiration
Status: Terminated | Type: Observational
Why Stopped: Recruitment rates too low to continue with the study
Sponsor: ProTiP Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: NB for HNC
Record Dates: First submitted 2015-04-23; First posted 2015-05-07 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-04

CONDITIONS: Aspiration; Laryngeal Cancer
Keywords: Dysphagia; Aspiration; Laryngeal cancer
MeSH Terms: conditions — Laryngeal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NewBreez: The study group is composed only of patients who have already opted to receive the NewBreez device as part of their routine care from their physician.
  Patients who have the device implanted, and consent to be part of the 12 week observational study, will be enrolled and have standard clinical parameters measured over the 12 week period as well as complete quality of life assessments in the form of patient questionnaires.
  Interventions: Device: NewBreez

INTERVENTIONS:
Device: NewBreez — Intralaryngeal prosthesis to protect the airways
  Other Names: Intralaryngeal Prosthesis

SUMMARY:
Laryngeal dysfunction is a problem that affects many patients after laryngeal cancer therapy (surgery or radio/chemotherapy). Laryngeal dysfunction is associated with higher incidences of aspiration and respiratory tract complications such as aspiration pneumonia. Current standard of care treatment to reduce the consequences of aspiration is often a tracheostomy which has its own risks and complications. The proposed study aims to describe the performance of a new CE marked medical implant, the NewBreez, in protecting the patient's airways from aspiration.

DETAILED DESCRIPTION:
Aspiration is associated with respiratory tract infections, reduced quality of life and increased mortality in patients. For chronic or unresolved aspiration, patients are often given a tracheostomy for safer breathing and greater protection of the airways from aspirated material. However tracheostomies are associated with risks and complications and do not give a 100% guarantee of aspiration protection to the patient. They also impact the quality of life in a negative way for many patients. The current study will evaluate the performance of a new intralaryngeal device for airway protection in a small group of patients who have chronic aspiration. The study will look at the overall performance of this device in preventing aspiration in this specific group of patients as well as determine any unforeseen risks of using this device in the identified group of patients. The outcomes will form the basis of future studies with larger groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* History of head and neck cancer
* Chronic aspiration
* Currently has a tracheostomy
* Patient is able to independently maintain their tracheostomy and cannula apparatus
* Patient meets the CE Mark indications and are not contraindicated for a NewBreez procedure.
* Anatomically compatible with the available sizes of NewBreez®
* 18 years of age or older
* Sufficient cognitive function to comply with the study and follow-up requirements
* Patient gives voluntary signed informed consent

Exclusion Criteria:

* Recurrent or present cancer in the previous 12 months
* Absent cough reflex
* Severely disrupted swallowing function e.g. severe neurological deficit, absent swallowing reflex, severe fixation of the larynx due to scarring with absent elevation of the larynx
* Upper esophageal sphincter not functional e.g. remains closed
* Cor Pulmonale / Pulmonary Heart Disease, or current lung infection
* Mouth opening less than 3.5cm
* Neck extension severely restricted hindering implantation of the device
* Contraindication to general anesthesia
* Severe hyperostosis (spondylophytes) of the cervical vertebrae causing dysphagia
* Severe (radiogenic) edema or damage of the mucosa of the upper aerodigestive tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients will primarily be from the department of Ear, Nose and Throat at the hospitals participating in the study. Secondary recruitment could also include associated clinics that treat patients with laryngeal dysfunction and aspiration, such as swallowing therapy clinics, speech language therapy clinics, and linguistics clinics.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schroeder, Dr. med., Principal Investigator — University of Luebeck

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- NewBreez: The study group is composed only of patients who have already opted to receive the NewBreez device as part of their routine care from their physician.
  Patients who have the device implanted, and consent to be part of the 12 week observational study, will be enrolled and have standard clinical parameters measured over the 12 week period as well as complete quality of life assessments in the form of patient questionnaires.
  NewBreez: Intralaryngeal prosthesis to protect the airways
Period: Overall Study
Arm/Group | NewBreez
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | NewBreez
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Per Patient of Number and Severity of Aspiration Events
Description: In patient change from baseline measurement of aspiration severity and frequency of events at weeks 1,4,8,and 12
Time Frame: 12 weeks
Population: First patient: Device was explanted within 48 hours after implantation - no Data could be collected Second Patient: Due to patient's non-compliance no data could be collected.Device was explanted within two weeks after implantation.
Arm/Group | NewBreez
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Reported Adverse Events
Description: Analysis of the reported system or procedure related adverse events using standard AE reporting form
Time Frame: at device implantation
Measure: Number; unit: adverse events
Arm/Group | NewBreez
Number analyzed (Participants) | 2
adverse events | 0

3. Secondary Outcome: Number of Reported Adverse Events
Description: Analysis of the the rate and severity of reported system or procedure related adverse events as a measure of safety of the device in this patient population over a 12 week period
Time Frame: 2 weeks
Measure: Number; unit: AE reported
Arm/Group | NewBreez
Number analyzed (Participants) | 2
AE reported | 2

4. Secondary Outcome: Number of Participants With an Increase of Greater Than 1 on the Heyse-Moore Score
Description: In patient change from baseline score of dyspnea using Heyse-Moore (Dyspnea)score:
  0 = None
  1. = Mild, some difficulty
  2. = Moderate Difficulty but can continue
  3. = Severe difficulty, cannot continue
Time Frame: 1 weeks
Population: Second enrolled patient did not reach the first data point, subj. was explanted prior first measurement.
Measure: Number; unit: participants
Arm/Group | NewBreez
Number analyzed (Participants) | 1
participants | 1

5. Other Pre Specified Outcome: Number of Participants With Reported Device Migration in the Larynx Post Implant
Description: In patient change from baseline position of the device in the larynx of each patient assessed by endoscopy and/or other clinically appropriate methods (CT or video fluoroscopy) and recorded in migration direction and distance (cm)
Time Frame: 1 weeks
Measure: Number; unit: participants
Arm/Group | NewBreez
Number analyzed (Participants) | 2
participants | 1

6. Other Pre Specified Outcome: Change From Baseline of Quality of Life (QoL) Score
Description: In patient QoL assessed at baseline and at 12 weeks using German standard QoL clinical questionnaire specifically for patients with swallowing dysfunction
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Reported Subjective Rating of Comfort of the Device in the Larynx
Description: In patient subjective measure (repeated) of pain score (1-10) and comfort level (questionnaire) at weeks 1,4,8,12
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: subject 1: 24 hours after receiving the NewBreez implant subject 2: 11 days after receiving the NewBreez implant
Arm/Group | NewBreez
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NewBreez (N=2)
aspiration (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NewBreez (N=2)
Device migration (Product Issues) | 1 (1) — device failed to remain in the intended location in the larynx

LIMITATIONS AND CAVEATS:
Very low recruitment achieved over all sites and early termination of the enrolled subjects gives insufficient data for any meaningful analysis of the product performance and safety in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No